CLINICAL TRIAL: NCT02682238
Title: A Multicenter, Randomized, Double-Blinded, Vehicle-Controlled Study to Evaluate the Safety and Local Tolerability of Topically Applied BBI-4000 (Sofpironium Bromide) 15% Gel in Subjects With Palmar Hyperhidrosis
Brief Title: A Safety, Tolerability and Preliminary Efficacy Study of BBI-4000 Gel in Subjects With Palmar Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI-4000-CL-202
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BBI-4000, 15% (Experimental): 15% BBI-4000 (sofpironium bromide) topical gel
  Interventions: Drug: BBI-4000, 15%
- Vehicle (Placebo Comparator): Vehicle (placebo) gel
  Interventions: Other: Vehicle gel

INTERVENTIONS:
Drug: BBI-4000, 15%
  Arms: BBI-4000, 15%
Other: Vehicle gel
  Other Names: Placebo gel
  Arms: Vehicle

SUMMARY:
To assess the safety and local tolerability of BBI-4000 15% gel compared with vehicle (placebo) when applied topically once daily in subjects with palmar hyperhidrosis.

DETAILED DESCRIPTION:
This is a Multicenter, Randomized, Double Blind, Vehicle-Controlled Study to Evaluate the Safety and Local Tolerability of Topically Applied BBI-4000 (Sofpironium Bromide) 15% Gel in Subjects with Palmar Hyperhidrosis.

Participating subjects will apply either BBI-4000 15% or vehicle gel topically to the palms of both hands once daily for 4 consecutive weeks. The 4 week treatment period will be followed by a 2 week follow-up period.

Safety and tolerability will be assessed through collection of vital signs, adverse events, assessment of local skin responses, ECG, UPT and blood sampling.

Efficacy will be assessed through gravimetric sweat assessments as well as through the Hyperhidrosis Disease Severity Scale (HDSS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary palmar hyperhidrosis
* HDSS of 3 or 4 at baseline
* Gravimetric test at baseline indicating at least 100 mg of sweat production at rest in each palm and a sum of at least 250 mg in both palms, in 5 minutes (room temperature)
* Symptoms of at least 6 months' duration
* Females of childbearing potential must agree to use a medically acceptable method of contraception while participating in the study

Exclusion Criteria:

* Any skin or subcutaneous tissue conditions of the palms, other than hyperhidrosis
* Prior use of any prohibited medication(s) or procedure(s) within specified timeframe for the treatment of palmar hyperhidrosis, including:

  1. Botulinum toxin to the palmar area within 9 months of baseline visit
  2. Iontophoresis within 30 days of baseline visit
  3. Palmar thermolysis, sympathectomy or surgical procedures of the palmar area any time in the past
  4. Serotonergic agonist within 30 days of baseline visit
  5. Any topical prescription treatment for hyperhidrosis within 30 days of baseline visit
  6. Any over-the-counter topical antiperspirant/deodorant within 7 days of baseline visit
* Use of anticholinergic agents within 30 days of baseline visit
* Any oral or topical homeopathic or herbal treatment within 30 days of baseline visit
* Use of any cholinergic drug within 30 days of baseline visit
* Use of any anti-anxiety and/or anti-depressant, amphetamine products or drugs with known anticholinergic side effects
* Hyperhidrosis secondary to any known cause
* Subjects with history of unstable type 1 or type 2 diabetes mellitus or thyroid disease, history of renal impairment, hepatic impairment, malignancy, glaucoma, intestinal obstructive or motility disease, obstructive uropathy, myasthenia gravis, benign prostatic hyperplasia (BPH), neurological conditions, psychiatric conditions, Sjögren's syndrome, Sicca syndrome, or cardiac abnormalities that may alter normal sweat production or may be exacerbated by the use of anticholinergics.
* Subjects with known hypersensitivity to glycopyrrolate, anticholinergics, or any of the components of the topical formulation.
* Pregnant or lactating women.
* Use of an investigational drug within 30 days prior to the baseline visit.
* Any major illness within 30 days before the screening examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2016-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - TCR Medical Corporation, San Diego, California
  - International Dermatology Research, Inc., Miami, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - Saint Louis University Dermatology, St Louis, Missouri
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- BBI-4000 (Sofpironium Bromide) Gel, 15%: BBI-4000 (sofpironium bromide) gel, 15%, one-pump applied to each palm nightly
- Vehicle Gel: Vehicle (placebo) gel, one-pump applied to each palm nightly
Period: Overall Study
Arm/Group | BBI-4000 (Sofpironium Bromide) Gel, 15% | Vehicle Gel
Started | 25 | 25
Completed | 22 | 21
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance with Study Drug | 1 | 0
Not completed — Non-compliance with Protocol | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- BBI-4000, 15%: 15% BBI-4000 (sofpironium bromide) topical gel
  BBI-4000, 15%
- Vehicle: Vehicle (placebo) gel
  Vehicle gel
- Total: Total of all reporting groups
Arm/Group | BBI-4000, 15% | Vehicle | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (30) | 30.5 (28) | 31.1 (30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 17 | 21 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events by Severity
Description: Each subject counted only once. Severity was rated Mild, Moderate or Severe.
Time Frame: Baseline visit-Day 42 End of Participation
Population: Participants receiving applying at least one dose of investigational treatment
Measure: Number; unit: Number of Events by Severity
Groups:
- BBI-4000 Gel, 15%: BBI-4000 Sofpironium bromide gel,15% applied once to each palm daily for 28 days
- Vehicle Gel (Placebo): Vehicle gel (placebo), applied once to each palm daily for 28 days
Arm/Group | BBI-4000 Gel, 15% | Vehicle Gel (Placebo)
Number analyzed (Participants) | 24 | 25
Number of Events by Severity
  Mild | 14 | 4
  Moderate | 3 | 0
  Severe | 0 | 0

2. Secondary Outcome: Proportion of Randomized Subjects Achieving a 1-grade & 2-grade Decrease in Hyperhidrosis Disease Severity Scale (HDSS) From Baseline to Day 29
Description: HDSS assessment included a progressive hyperhidrosis severity scale, in which participants would rate the severity of their palmar hyperhidrosis for the past week with one of the following: 1-My sweating is never noticeable and never interfered with my daily activities; 2-My sweating is tolerable but sometimes interferes with my daily activities; 3-My sweating is barely tolerable and frequently interferes with my daily activities; 4-My sweating is intolerable and always interferes with my daily activities
Time Frame: Baseline to Day 29 (End of Treatment) Visit
Population: Randomized participants who provided HDSS scores: baseline and day 29
Measure: Count of Participants; unit: Participants
Groups:
- BBI-4000 (Sofpironium Bromide) Gel, 15%: BBI-4000 Sofpironium bromide gel, 15%, applied once to each palm daily for 28 days
Arm/Group | BBI-4000 (Sofpironium Bromide) Gel, 15% | Vehicle Gel (Placebo)
Number analyzed (Participants) | 22 | 23
Participants
  Proportion of Subjects with at least 1-Point Decrease : No | 8 | 6
  Proportion of Subjects with at least 1-Point Decrease : Yes | 14 | 17
  Proportion of Subjects with at least 2-Point Decrease : No | 20 | 21
  Proportion of Subjects with at least 2-Point Decrease : Yes | 2 | 2

3. Secondary Outcome: Absolute Change (Day 29 - Baseline) in Palmar Gravimetrically Measured Sweat Production (GMSP) (mg) by Treatment Arm.
Description: Individual Right and left palm gravimetric measured sweat production results (mg) were combined per participant at Baseline and Day 29 time points. Mean averages of individual absolute GMSP changes (Day 29 Combined GMSP-Baseline Combined GMSP) were compared between the two treatment arms.
Time Frame: Baseline-Day 29 Participation
Population: Randomized participants (to one of two treatment arms) who provided Gravimetrically Measured Sweat Production (GMSP) results (Right and Left Palms) Baseline and day 29
Measure: Mean (Standard Deviation); unit: mg
Units Other Than Participants: Palm
Groups:
- Vehicle Gel (Placebo): Vehicle (placebo) gel, applied once to each palm daily for 28 days
Arm/Group | BBI-4000 (Sofpironium Bromide) Gel, 15% | Vehicle Gel (Placebo)
Number analyzed (Participants) | 22 | 23
Number analyzed (Palm) | 88 | 92
mg | -91.38 (385.12) | -156.62 (367.69)

4. Secondary Outcome: Comparison of Number Subjects Achieving a Minimum of 50% Reduction in Gravimetrically Measured Sweat Production Day 29-baseline Among Both Treatment Arms
Description: Visit combined sweat production (mg) was calculated by combining individual right and left palm gravimetric sweat production results (mg) at Baseline and Day 29 time points. Resulting difference was calculated by: Day 29 Combined GMSP - Baseline Combined GMSP. Percent reduction in sweat production was calculated by: ((Resulting difference GMSP score (mg)) / Baseline GMSP score (mg) x 100). The number of subjects who achieved ≥ 50% reduction in sweat production (YES) were reported, along with the proportion=number of subjects who achieved ≥ 50% reduction in sweat production / total number of subjects providing baseline and day 29 results x 100. The number of subjects who achieved < 50% reduction in sweat production (NO) were reported, along with the proportion=number of subjects who achieved < 50% reduction in sweat production / total number of subjects providing baseline and day 29 results x 100.
Time Frame: Baseline through day 29 (End of Treatment)
Population: Randomized participants completing baseline through day 29 (End of Treatment) activities. Note: For this analysis, number analyzed includes 22 (gel, 15%) and 23 (Placebo) participants, and 22 (gel, 15%) and 23 (Placebo) participants' % reduction in sweat production for analysis.
Measure: Number; unit: participants
Units Other Than Participants: Palm
Groups:
- BBI-4000 Sofpironium Bromide Gel, 15%: BBI-4000 Sofpironium bromide gel, 15%, applied once to each palm daily for 28 days
- Vehicle Gel, (Placebo): Vehicle (placebo) gel, applied once to each palm daily for 28 days
Arm/Group | BBI-4000 Sofpironium Bromide Gel, 15% | Vehicle Gel, (Placebo)
Number analyzed (Participants) | 22 | 23
Number analyzed (Palm) | 88 | 92
participants
  The number of subjects who achieved < 50% reduction in sweat production (NO) | 18 | 18
  The number of subjects who achieved ≥ 50% reduction in sweat production (YES) | 4 | 5

5. Secondary Outcome: The Percent Change (%) Day 29 Combined GMSP From Baseline Combined GMSP Gravimetrically Measured Sweat Production (GMSP) in Combined (Right and Left) Palms.
Description: Individual Right and left palm gravimetric sweat production (GMSP) results (mg) were combined per participant at Baseline and Day 29 time points. Mean averages of individual percent change were compared between the two treatment arms. Individual % Change vs. Baseline was determined by: [(D29 Right palm GMSP + D29 Left palm GMSP)-(Baseline Right palm GMSP + Baseline Left palm GMSP)]/(Baseline Right palm GMSP + Baseline Left palm GMSP)]
Time Frame: Baseline-Day 29 End of Treatment
Population: Participants applying at least one dose of investigational treatment to each palm and providing both right & left palm GMSP results at baseline and day 29. Combined GMSP results were determined by adding GMSP Left Palm + GMSP Right Palm results.
Measure: Mean (Standard Deviation); unit: percentage of change
Units Other Than Participants: Palm
Groups:
- BBI-4000 (Sobpironium Bromide) Gel, 15%: BBI-4000 (sofpironium bromide) topical gel, 15%, one-pump (per palm) applied to each palm once at night
- Vehicle Gel: Vehicle (placebo) gel, one-pump (per palm) applied to each palm once at night
Arm/Group | BBI-4000 (Sobpironium Bromide) Gel, 15% | Vehicle Gel
Number analyzed (Participants) | 22 | 23
Number analyzed (Palm) | 88 | 92
percentage of change | -10.56 (52.61) | -15.76 (45.05)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of consent signature (screening period was ≤ 30 days), baseline, day 29 (end of treatment), through to day 42 (± 3 days) (safety follow-up); overall duration of adverse collection for each participant could be up to 75 days
Description: Subjects with Treatment Emergent Adverse Events (TEAEs). The Safety population (N=49) included all subjects enrolled in the study who were dispensed and applied study drug at least once. One subject was excluded from the Safety population because the subject did not apply any study drug.
Groups:
- BBI-4000, 15%: 15% BBI-4000 (sofpironium bromide) topical gel, one pump applied to each palm nightly
- Vehicle: Vehicle (placebo) gel, one pump applied to each palm nightly
Arm/Group | BBI-4000, 15% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 8/24 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BBI-4000, 15% (N=24) | Vehicle (N=25)
Application Site Dermatitis (General disorders) | 2 | 0
Application Site Hyperaesthesia (General disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 0
Mydriasis (Eye disorders) | 2 | 0
Vision Blurred (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Application Site Eczema (General disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement terms prioritized a multi-center publication at the study end. Should such a publication not be completed, an investigator right to individually publish results of his/her study (limited to his/her site data) was included, if for purely scientific or educational purposes; not for any commercial purposes. PI(s) were to submit draft materials to the Sponsor 60 days prior to Investigator release of individual abstract or manuscript. Additional disclosure restrictions and terms applied .